CLINICAL TRIAL: NCT00211393
Title: A Pilot Study of The Treatment of Central Serous Chorioretinopathy With Ketoconazole.
Acronym: CSC/Keto
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: LuEsther T. Mertz Retinal Research Center (Other)
Responsible Party: Principal Investigator, Joan, K. Bailey Freund, M.D., Manhattan Eye, Ear & Throat Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M00.013
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Central Serous Chorioretinopathy
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: ketoconazole (Experimental): Drug: ketoconazole
  Other Names:
  ketoconazole
  600mg. /day for 6 weeks
  --------------------------------------------------------------------------------
  Interventions: Drug: ketoconazole

INTERVENTIONS:
Drug: ketoconazole — 600mg. /day for 6 weeks

SUMMARY:
The purpose of this study is to determine the effect of an adrenocorticoid antagonist (ketoconazole), 600 mg per day for 4 weeks, in the treatment of patients with central serous chorioretinopathy (CSC).

DETAILED DESCRIPTION:
A complete ophthalmic evaluation and tests: autofluorescence and Fluorescein angiography, Color Fundus Photography, OCT, including liver and adrenal functions and pregnancy test, if applicable will be done on the screening visit. If the patient is eligible, the patient will be started on ketoconazole 600 mg per day by mouth for the following next 6 weeks. The patient will be rechecked at weeks 5-6, 10,14 and 18. During all these visits a complete ophthalmic examination autofluorescence, OCT, and color fundus photographs will be done.

Repeat Liver and Adrenal function tests will be done at weeks 5-6 and 10 visits.

On the exit visit, all the ophthalmic tests and procedures on the baseline visit will be done. Adverse events, and concomitant medications and treatments will be reported on all visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 60 years
2. Must have clinical signs of CSC with leakage from the level of the RPE during fluorescein angiography and neurosensory detachment documented by optical coherence tomography (OCT).
3. Be able to return for all study visits for 3 months' duration.
4. Be able to provide written informed consent
5. Must have sufficiently clear media to allow for adequate fundus photography

Exclusion Criteria:

1. Have choroidal neovascularization.
2. Have any evidence of clinically significant intraocular inflammation, angioid streaks, presumed ocular histoplasmosis syndrome, or other precursor of choroidal neovascularization.
3. Have additional eye disease that compromises the visual acuity of the study eye.
4. Are receiving any systemic steroid therapy
5. Have any significant medical history
6. Have a history of severe hypersensitivity reaction to any of the dyes or the drug used in the study.
7. Have any history of ocular conditions that may mimic CSC
8. Are pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Visual acuity (ETDRS) after 6 weeks of treatment | 18 weeks

SECONDARY OUTCOMES:
Changes in the choroidal vascular pattern as observed on FA and changes at the posterior pole as measured with optical coherence tomography | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: K. Bailey Freund, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States